CLINICAL TRIAL: NCT07063420
Title: Patient Centered Multi-Agent Decision Support System (PCM-DSS) for Healthcare Providers: A Pilot Study
Brief Title: Patient Centered Multi-Agent Decision Support System (PCM-DSS) for Healthcare Providers
Acronym: TREAT2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Chernavvsky, MD (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor-Investigator, Daniel Chernavvsky, MD, Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 302621
Record Dates: First submitted 2025-06-17; First posted 2025-07-14 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Patient Centered Multi-Agent Decision Support System (PCM-DSS); Continuous Glucose Monitor (CGM); Insulin pen
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM + Patient Centered Multi-Agent Decision Support System (PCM-DSS) (TREAT2) (Experimental): Participants will use their personal insulin pen and study continuous glucose monitor (CGM). Participants will adjust therapy guided by the study physician who receives the TREAT2D Report for a 16-week period. TREAT2D Report is generated by the Patient Centered Multi-Agent Decision Support System (PCM-DSS). Participant will then complete a 2-week Maintenance Phase where therapy established during the Intervention Phase will be maintained.
  Interventions: Other: Continuous Glucose Monitor (CGM) + Patient Centered Multi-Agent Decision Support System (PCM-DSS)
- CGM + Usual Care (Physician) (Placebo Comparator): Participants will use a study CGM and their personal insulin pen. They will have their insulin therapy guided by the study physician for a 16-week period. Participants will be contacted by study personnel as per standard care to adjust their therapy if needed. Participants will then complete a 2-week Maintenance Phase where therapy established during the Intervention Phase will be maintained.
  Interventions: Other: Continuous Glucose Monitor (CGM) + Usual Care

INTERVENTIONS:
Other: Continuous Glucose Monitor (CGM) + Patient Centered Multi-Agent Decision Support System (PCM-DSS) — Continuous Glucose Monitor (CGM) + Patient Centered Multi-Agent Decision Support System (PCM-DSS) PCM-DSS
  Arms: CGM + Patient Centered Multi-Agent Decision Support System (PCM-DSS) (TREAT2)
Other: Continuous Glucose Monitor (CGM) + Usual Care — Continuous Glucose Monitor (CGM) + Usual Care (Physician)
  Arms: CGM + Usual Care (Physician)

SUMMARY:
Decision Support System (Software) for multi antidiabetic drug therapy use in type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The purpose of this study is to test the safety and feasibility of using a patient centered decision support system (software) aim for healthcare providers to treat people with type 2 diabetes under multi antidiabetic drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 years old at time of consent.
2. Clinical diagnosis, based on investigator assessment, of type 2 diabetes for at least 6 months.
3. Hemoglobin A1c (HbA1c) ≥ 7.0%.
4. Currently using an approved long-acting insulin for at least 3 months (e.g., insulin glargine, insulin degludec).
5. Treated or about to be treated with multi-drug therapies for T2D.
6. If using a CGM, willingness to wear an additional study CGM during the duration of the study.
7. Access to the internet and willingness to upload data during the study as needed.
8. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females who self-report that they are of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.

Exclusion Criteria:

1. Currently using rapid insulin for at least three months (e.g., insulin aspart, insulin lispro, insulin regular).
2. Currently being treated for a seizure disorder.
3. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol, such as but not limited to, the following examples:

   1. Seizure disease
   2. Decompensated cardiac disease
4. Inpatient psychiatric treatment in the past 6 months
5. Presence of a known adrenal disorder
6. Currently pregnant or intent to become pregnant during the trial.
7. Anticipated surgical, interventional procedures or prolonged periods of fasting during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | 22 weeks
  Measured by improved glycemic control (HbA1c change and CGM-derived metrics).

OTHER OUTCOMES:
Patient satisfaction | 22 weeks
  Patient satisfaction which will be assessed through Diabetes Distress Scale Survey (DDS) questionnaire, measured after Screening and at End of Study, and the Participant Satisfaction Survey (PSS) measured at End of Study. DDS asks the participant to consider the degree distress they felt to 17 items during the past month. PSS is six questions asking the participant about the experience in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Nass, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after the publication of the manuscript.
Access Criteria: The Data Sharing Agreements will be formulated by the study team